CLINICAL TRIAL: NCT07246278
Title: Evaluating Safety and Efficacy of Celecoxib in Patients With PD.
Brief Title: Celecoxib in Parkinson Disease as Adjuvant Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5478
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): control group ( levo-dopa group, n =40 ) who will receive levo-dopa/carbidopa (125/12.5) mg three times daily for 6 months.
  Interventions: Drug: Levodopa Carbidopa
- Celecoxib group (Active Comparator): will receive levo-dopa/carbidopa (125/12.5) mg three times daily plus celecoxib 200 mg once daily.
  Interventions: Drug: Levodopa Carbidopa; Drug: Celecoxib 200mg

INTERVENTIONS:
Drug: Levodopa Carbidopa — Carbidopa/levodopa is the combination of the two medications carbidopa and levodopa. It is primarily used to manage the symptoms of Parkinson's disease
Drug: Celecoxib 200mg — Celecoxib, is a selective cyclooxygenase-2 inhibitor. Prostaglandins (PG) are produced from arachidonic acid by the constitutively expressed cyclooxygenase-1(COX-1)
  Arms: Celecoxib group

SUMMARY:
Parkinson's disease (PD) is a chronic neurodegenerative disease clinically characterized by bradykinesia, hypokinesia, rigidity, resting tremor, and postural instability. These motor manifestations are attributed to the degeneration and selective loss of dopaminergic neurons in the substantia nigra pars compacta (SNpc), leading to a dopamine (DA) deficiency in the striatum. Neuroinflammation is considered one of the most important factors contributing critically to pathophysiology of PD . Recently, high mobility group box-1 (HMGB1) protein has been encoded as a potential inflammatory biomarker in PD

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both male and female will be included.
* Patients diagnosed with PD according to Unified Parkinson's Disease Rating Scale.

Exclusion Criteria:

* Breast feeding
* Patients with significant liver and kidney function abnormalities.
* Alcohol and / or drug abusers.
* Patients with known allergy to the study medications
* Patients with known allergy to sulfonamides (cross hypersensitivity with celecoxib).
* Pregnant women and women with planned pregnancy.
* Patients who are currently using other anti-inflammatory drugs.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
change in the Unified Parkinson's Disease Rating Scale | 6 months
  - Change From Baseline for Unified Parkinson's Disease Rating Scale (UPDRS) Total Score

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt